CLINICAL TRIAL: NCT03701204
Title: Integrating Contingency Management Into Routine Care for Alcohol Use Disorder
Brief Title: Contingency Management for Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DynamiCare Health (Industry)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Eric Gastfriend, Principal Investigator, DynamiCare Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DCH001
Record Dates: First submitted 2018-10-07; First posted 2018-10-09 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DynamiCare Rewards (Experimental): The study will test the feasibility/acceptability and efficacy of DynamiCare Rewards™. DynamiCare Rewards is an iOS/Android app which automates Contingency Management (CM) to help the patient self-monitor and focus attention on his/her behavioral goals (i.e., abstinence) for alcohol or other substance use disorders.
  Interventions: Behavioral: DynamiCare Rewards
- Control (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: DynamiCare Rewards — Participants assigned to the DynamiCare Rewards group will receive the following:
  1. App on their smartphone
  2. Substance Testing Devices: BACTrack Mobile Pro - submits BAC results directly to smartphone via Bluetooth and Saliva Test Kits.
  3. Next Step debit card to receive financial incentives
  4. Participant will be prompted via the app to conduct breathalyzer/saliva tests, using the devices camera to take "selfie" photo/videos to prevent cheating.
  5. Negative tests result in participant receiving electronic virtual "coins", which can be transferred from reserve account (reserve account inaccessible to participant) to the spendable Next Step debit card.
  6. The amount of coins and funds are available on a progressive variable reward schedule.
  Arms: DynamiCare Rewards

SUMMARY:
Randomized pilot study of a device (smartphone app) that poses non-significant risk to participants and is exempt from Investigational Device Exemption regulations [21 Code of Federal Regulations 812.2(c)

DETAILED DESCRIPTION:
To test the feasibility/acceptability and efficacy of a minimum viable product (MVP) of a smartphone app for patients with alcohol use disorder who are in active treatment and recovery to perform self-tracking of their recovery behavior (e.g., abstinence) and focus on their motivation to maintain their desired health behaviors (i.e., abstinence).

ELIGIBILITY:
Inclusion Criteria:

Participants in the pilot study will be 60 new intakes to Gosnold's outpatient Substance Use Disorder (SUD) program who:

* are >18 years old;
* meet DSM-5 criteria for current (past year) alcohol use disorder, at least moderate severity;
* identify alcohol as the primary drug problem;
* Currently use alcohol (past 7 days) or have been in treatment 14 days or less and used alcohol within 7 days of treatment entry;
* have and use an Android or iOS smartphone with acceptable
* capability;
* are willing to participate in home testing and use of the smartphone,
* speak and read the English language adequately to understand smartphone commands and responses and
* are willing to be randomly assigned to receive treatment with or without the smartphone app as an added feature.

Exclusion Criteria:

• Participants must not currently be suicidal or actively psychotic, by clinician judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2019-08-21 (Actual)

PRIMARY OUTCOMES:
Percent of participants abstinent from alcohol at each monthly assessment time point (negative urine test and self-report of no use in past 30 days) | 12-week intervention period
  The pilot efficacy study will utilize alcohol abstinence at each assessment time point as the primary outcome. This is defined as a negative ethyl glucuronide urine test (witnessed) at the monthly assessment time points and self-report of no alcohol use in the past 30 days.

SECONDARY OUTCOMES:
Percent of participants abstinent from all drugs at each monthly assessment time point (negative urine test and self-report of no use in past 30 days) | 12-week intervention period
  Groups will be compared using Generalized Estimating Equation (GEE) analysis on the percent of participants abstinent over time at each time point.
Longest continuous period of abstinence from alcohol and from drugs and alcohol | 12-week intervention period
  Groups will be compared using GEE analysis on the percent of participants abstinent over time at each time point.
Retention in treatment | 12-week intervention period
  Groups will be compared on the number of days retained in treatment according to the site's Electronic Health Record data, and also on the graduation rate from treatment vs. leaving against medical advice.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Gastfriend, MBA, Principal Investigator — DynamiCare Health
Locations (2):
- United States (2):
  - Gosnold on Cape Cod, Centerville, Massachusetts
  - Gosnold, Falmouth, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided
We intend to make participant data available by request as long as it is unidentifiable.